CLINICAL TRIAL: NCT02475811
Title: The Role of 3D Ultrasonography Fetal Lung Volume Measurement in the Prediction of Neonatal Respiratory Function Outcome
Brief Title: 3D Ultrasonography Fetal Lung Volume Measurement and Neonatal Respiratory Function
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, Assistant professor, Cairo University
Other Study IDs: 137
Record Dates: First submitted 2015-06-15; First posted 2015-06-19 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Neonatal Respiratory Function
Keywords: 3D ultrasonography; fetal Lung Volume; neonatal respiratory function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: 3D ultrasonography — The angle of volume sampling varied throughout gestational age with a maximum limit of 75° in the third trimester. After scanning the volume, multiplanar imaging in the 3 orthogonal ultrasonographic sections was analyzed to reconstruct the 3D ultrasound image. Before its volume was analyzed, each lung was carefully identified on the 3 orthogonal multiplanar imaging sections. We used the rotational technique that entails the VOCAL imaging program to measure lung volume. A transverse section of the multiplanar imaging was chosen as the reference image for volume analyses

SUMMARY:
One hundred healthy women with singleton pregnancies in the 1st stage of labor will be included in the study, divided into two groups; Group A (n: 50 - women pregnant ± 34-37 weeks) & Group B (n: 50 - women pregnant ± 37+1-40 weeks). A 3D volume model of the right fetal lung is generated & lung volume is calculated using VOCAL software. After child birth, neonatal respiratory functions will be assessed using APGAR score at (1, 5 and 10 min) together with occurrence of RDS and the further need for NICU admission and respiratory support measurements.

DETAILED DESCRIPTION:
One hundred healthy women with singleton pregnancies presented in the 1st stage of labour will beincluded in the study. Participants will be divided into two groups; Group A (n: 50 - women pregnant ± 34-37 weeks gestation) & Group B (n: 50 - women pregnant ± 37+1-40 weeks gestation). Gestational age (GA) is established by menstrual dates then confirmed by obstetric ultrasound.

For both groups, full history will be taken including the receiving of antenatal steroids followed by general, abdominal & pelvic examination to confirm the stage of labour & to exclude the presence of rupture of membranes. Obstetric ultrasound will be done to confirm GA, assess amniotic fluid index (AFI) & to exclude fetal anomalies. Fetal lung volume (FLV) measured using Voluson 730 Expert ultrasonography machine (GE Healthcare Austria GmbH, Seoul, Korea) equipped with a 4- to 8- MHz transabdominal transducer for 3-dimensional (3D) volume scanning. A single examiner will perform all ultrasound examinations with the following technique; a transverse section of the fetal thorax at the level of the 4-chamber view, with the fetal heart proximal to the transducer, was identified by 2-dimensional ultrasonography, and the volume box will be adjusted to scan the entire fetal thorax. The maximum resolution will be adjusted. The angle of volume sampling varied throughout gestational age with a maximum limit of 75° in the third trimester. After scanning the volume, multiplanar imaging in the 3 orthogonal ultrasonographic sections will be analyzed to reconstruct the 3D ultrasound image. Before its volume was analyzed, each lung was carefully identified on the 3 orthogonal multiplanar imaging sections. The investigators will use the rotational technique that entails the VOCAL imaging program to measure lung volume. A transverse section of the multiplanar imaging will be chosen as the reference image for volume analyses (Figure 1). Right lung volume will be measured by a series of area tracing of the studied lung after serial rotations of 30° (6 times; Figures 2 and 3). Reviewing parallel slices executed through the whole lung in the 3 perpendicular planes allowed us to check the adequacy of our rotational area tracing approach. Right lung volume was automatically measured and plotted against gestational age, taking about 2 minutes to estimate the lung volume. After child birth, neonatal respiratory functions will be assessed using APGAR score at (1, 5 and 10 min) together with occurrence of RDS and the further need for neonatal ICU admission and respiratory support measurements.

ELIGIBILITY:
Inclusion Criteria:

* One hundred healthy women with singleton pregnancies presented in the 1st stage of labour were included in the study. Participants were divided into two groups; Group A (n: 50 - women pregnant ± 34-37 weeks gestation) & Group B (n: 50 - women pregnant ± 37+1-40 weeks gestation). Gestational age (GA) is established by menstrual dates then confirmed by obstetric ultrasound

Exclusion Criteria:

* Exclusion criteria include the maternal administration of respiratory depressants within 2 hours from the delivery of the fetus (e. g., opioid analgesic & general anesthesia upon doing CS) or oligohydramnios (amniotic fluid index < 5th centile), rupture of membranes, the presence of fetal malformations (chest, heart or abdominal) or abnormal fetal growth (defined as: estimated fetal weight < 5th centile or > 95th centile and/or abdominal circumference < 5th centile or > 95th centile). Also, women with a cardiac pacemaker were excluded (as the transmitter necessary for the lung volume measurements could disturb the function of the pacemaker).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: One hundred healthy women with singleton pregnancies presented in the 1st stage of labour
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Apgar score | 1 minute after delivery

SECONDARY OUTCOMES:
Neonatal ICU admission | 24 hour after delivery
Apgar score | 5 minutes after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Maged, Principal Investigator — Kasr Alainy medical school
Locations (1):
- Kasr Alainy medical school, Cairo, Cairo Governorate, Egypt